CLINICAL TRIAL: NCT03278249
Title: Feasibility Study of Modified Atkins Ketogenic Diet in the Treatment of Newly Diagnosed Malignant Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Rekha Chaudhary, Associate Professor of Medicine, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-BRAIN-16-01
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma
Keywords: brain tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Atkins Ketogenic Diet (Experimental): Modified Atkins Ketogenic Diet in combination with Temodar and Radiation
  Interventions: Other: Modified Atkins Ketogenic Diet

INTERVENTIONS:
Other: Modified Atkins Ketogenic Diet — Less than 20 grams of carbohydrates per day

SUMMARY:
The purpose of this research study is to see if people can produce ketones in their blood with the modified Atkins diet. Modified Atkins diet is a diet that produces ketones in your blood by restricting carbohydrates to <20 grams per day. Ketones are substances that are produced in the blood when fat is being broken down. Ketones may help radiation work better and may starve your tumor because it is thought that some brain tumors can not use ketones to grow and can only use sugar or glucose to grow.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary malignant glioma, Grade III or IV
* No uncontrolled infection or other active malignancy or chronic systemic immune therapy.
* ECOG performance status < 3.
* Life expectancy > three months.
* Adequate labs

Exclusion Criteria:

* Diagnosis of genetic disorder of fat metabolism.
* Type 2 diabetes diagnosed with a hemoglobin A1C > 6.4
* Allergic to dairy or lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Chaudhary, MD, Principal Investigator — University of Cincinnati
Locations (1):
- UC Health, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified Atkins Ketogenic Diet
Started | 12
Completed | 9
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Modified Atkins Ketogenic Diet
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ketosis
Description: Ketosis measured by serum beta-hydroxybuterate. Ketosis is defined as having serum beta-hydroxybuterate (BHB) at > 0.05 mM. Participants' BHB levels were assessed at 6 weeks after starting the study. The number of participants who had BHB at > 0.05 mM were considered to have entered into ketosis. 9 of 9 participants met this criteria.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Atkins Ketogenic Diet
Number analyzed (Participants) | 9
Participants | 9

2. Secondary Outcome: Number of Participants With Progression Free Survival
Description: Progression Free Survival (PFS) is defined as the percentage of patients without progression at 6 months. Progression will be evaluated via Radiographic Assessment in Neuro-oncology (RANO) criteria: >5 mm increase in maximal diameter, as well as ≥ 25% increase in the sum of the products of the progressing.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Atkins Ketogenic Diet
Number analyzed (Participants) | 9
Participants | 6

3. Secondary Outcome: Assessment of Survival
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Atkins Ketogenic Diet
Number analyzed (Participants) | 9
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed for 2-3 months after pre-treatment visit 1, All-Cause Mortality monitored/assessed for up to 2 years
Description: The definitions do not differ from clinicaltrials.gov's definitions.
Arm/Group | Modified Atkins Ketogenic Diet
All-Cause Mortality (participants affected / at risk) | 3/9
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Atkins Ketogenic Diet (N=9)
Memory impairment (Nervous system disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Infection with unknown ANC - Wound (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Investigations, please specify (Investigations) | 1 (1)
Leukocytes (total WBC) (Investigations) | 1 (1)
Lymphatics - Other (Specify, __) (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1)
Platelets (Investigations) | 1 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Atkins Ketogenic Diet (N=9)
Allergic reaction (Immune system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Dizziness (Nervous system disorders) | 3 (3)
Edema: head and neck (General disorders) | 1 (1)
Edema: limb (General disorders) | 2 (2)
Fatigue (General disorders) | 7 (8)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2)
Hearing (Ear and labyrinth disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Investigations) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 2 (6)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extraocular (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-upper (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Facial (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Ocular (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Neurology - Other (Specify, __) (Nervous system disorders) | 2 (3)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (3)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1)
Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Head/headache (Nervous system disorders) | 1 (1)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Photosensitivity (Eye disorders) | 1 (2)
Platelets (Investigations) | 1 (1)
Potassium, serum-low (hypokalemia) (Investigations) | 2 (3)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 4 (4)
Rigors/chills (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Skin (cellulitis) (Infections and infestations) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Syndromes - Other (Specify, __) (General disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Urinary tract NOS (Infections and infestations) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 2 (3)
Wound (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT03278249/Prot_SAP_000.pdf